CLINICAL TRIAL: NCT01496625
Title: NEI Intramural Biorepository for Retinal Diseases
Brief Title: National Eye Institute Biorepository for Retinal Diseases
Status: Recruiting | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120042; 12-EI-0042
Record Dates: First submitted 2011-12-17; First posted 2011-12-21 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-10-06

CONDITIONS: Age-Related Macular Degeneration; Diabetic Retinopathy; Von Hippel-Lindau Syndrome; Retinal Disease; Retinal Vein Occlusion
Keywords: Biological Specimens; Retinal Disease; Diabetic Retinopathy; Phenotype-Genotype correlation; Age-Related Macular Degeneration (AMD); Natural History; AMD; Healthy Volunteer; HV
MeSH Terms: conditions — Macular Degeneration; Diabetic Retinopathy; von Hippel-Lindau Disease; Retinal Diseases; Retinal Vein Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Participants with age-related macular degeneration (AMD), diabetic retinopathy, and other retinal diseases.
- Cohort 2: Participants without any retinal diseases.

SUMMARY:
Background:

- To understand diseases of the retina and the eye, information is needed about people with and without such diseases. Researchers want to study these people and follow them over time. They also want to study body tissues and blood to understand the nature of eye disease. Studying genes, cells, and tissues may help them understand why some people get eye problems and others do not, or why some people respond to treatment while others do not. Researchers want to collect physical samples and personal data to develop a National Eye Institute database.

Objectives:

- To collect health information and blood and tissue samples from people with and without eye diseases, to be used in research studies.

Eligibility:

* Individuals at least 2 years of age with different types of eye disease.
* Healthy volunteers with no history of eye disease.

Design:

* Participants may be recruited from National Eye Institute studies or may be referred from other sources.
* Participants will be screened with a physical exam and medical history. They will also have a full eye exam. Questions will be asked about family medical history, especially about eye disease.
* Blood samples will be collected. Other samples, such as saliva, tears, hair, stool, and urine, may be collected as needed. Adult participants may also provide a skin sample.
* Tissue or fluid from eye collected as part of eye care or treatment may also be added to the database.
* No treatment will be provided as part of this study.

DETAILED DESCRIPTION:
This protocol establishes a clinical database and biospecimen repository for potential use in subsequent research projects approved by the NIH IRB, such as the identification of novel factors relevant to the pathogenesis, progression, and response to treatment of a variety of retinal conditions, particularly age-related macular degeneration (AMD) and diabetic retinopathy and their associated systemic correlates of disease.

Objectives: This protocol provides for standardized collection of longitudinal clinical data and for serial collection, processing, and storage of a variety of biospecimens. The clinical data set and biospecimen repository may be used in subsequent potential research studies for purposes including identification of novel genetic factors, biomarkers, and experimental models associated with pathogenesis, progression, and response to treatment for various conditions of the retina and their associated systemic correlates of disease.

Study Population: We plan to accrue up to 200 participants with AMD, 125 participants with diabetic retinopathy, 200 participants with other retinal diseases, and 125 participants without any retinal disease. A total of up to 650 participants may be enrolled.

Design: This protocol is designed around prospective observation of multiple retinal diseases and suitable controls incorporating:

Defined testing and ocular imaging on a standardized follow-up schedule; and

Collection of biospecimens for research purposes for which sampling does not incur more than minimal risk to participants.

Outcome Measures: Potential outcome measures for subsequent studies using this data set may include the interaction of key parameters of phenotype (such as visual acuity and retinal features on ocular imaging) with genetic variants and other biomarkers identified from biospecimens, and the characterization of new experimental models of eye health and disease.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants will be eligible if they:

* Have the ability to understand and sign an informed consent or have a parent/legal guardian to do so if they are minor children.
* Manifest diagnosed or undiagnosed retinal disease(s), or could serve as an unaffected control suitable for comparison to participants with various retinal diseases, particularly AMD and diabetic retinopathy (taking into account matching factors such as age and past ocular history).

EXCLUSION CRITERIA:

Participants will not be eligible if they:

* Are unable or unwilling to give informed consent that includes collection and study of at least one peripheral blood sample.
* Are unable or unwilling to give informed consent that includes use of NIH medical records and clinical samples for research.
* Have a systemic disease that compromises the ability to provide adequate ophthalmologic examination or treatment.

Ages: 2 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study accrual goal is up to 200 participants with AMD, 125 participants with diabetic retinopathy, 200 participants with other retinal diseases, and 125 participants without any retinal disease. A total of up to 650 participants may be enrolled. Participants may enroll in this study after referral by a medical practitioner in the private sector, or by another clinic, hospital, or medical institution. Participants may enroll in this study concurrently with another NEI or NIH protocol, or following completion of another study. Self-referral will be permitted. Advertisements will not be used.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2012-06-18 (Actual)

PRIMARY OUTCOMES:
The intent is to collect data on a variety of phenotypic parameters and to store biospecimens in a manner that permits a broad array of potential testing and experimentation in the future. | Ongoing
  In subsequent potential studies (dependent on separate IRB approval in each case), the outcome measures of the clinical data and samples from this protocol might include: (i) key parameters of phenotype from ophthalmic evaluation, such as visual acuity and aspects of ocular disease status documented by fundus imaging modalities like color photography, autofluorescence photography, and optical coherence tomography (OCT); (ii) other biomarkers identified from biospecimens.

CONTACTS AND LOCATIONS:
Overall Officials: Tiarnan DL Keenan, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
At this point it is undecided whether IPD will be shared.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2012-EI-0042.html